CLINICAL TRIAL: NCT01657903
Title: A Placebo Controlled Study to Evaluate the Effectiveness of Experimental Foaming Gel Toothpastes Using an In-situ Erosion Remineralization Model
Brief Title: Evaluation of Efficacy of Experimental Gel to Foam Dentifrices in Dental Erosion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Z6961385
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2014-07

CONDITIONS: Dental Erosion; Acid Wear
MeSH Terms: conditions — Tooth Erosion | interventions — Sodium Fluoride; potassium nitrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- NaF/KNO3 toothpaste, Low RDA (Experimental): Participants to brush with 1.5 g of low RDA gel to foam toothpaste containing 1450 ppm F - EU level as NaF. All study treatments contain 5% weight by weight (w/w) KNO3.
  Interventions: Drug: Sodium Fluoride; Drug: Potassium nitrate
- NaF/KNO3 toothpaste, Medium RDA (Experimental): Participants to brush with 1.5 g of medium RDA gel to foam toothpaste containing 1450 ppm F - EU level as NaF. All study treatments contain 5% w/w KNO3.
  Interventions: Drug: Sodium Fluoride; Drug: Potassium nitrate
- NaF/KNO3 toothpaste (Active Comparator): Participants to brush with 1.5 g of NaF/KNO3 toothpaste containing 1450 ppm F - EU level as NaF. All study treatments contain 5% w/w KNO3.
  Interventions: Drug: Sodium Fluoride; Drug: Potassium nitrate
- No fluoride/KNO3 toothpaste (Placebo Comparator): Participants to brush with a fluoride free toothpaste (0 ppmF). All study treatments contain 5% w/w KNO3.
  Interventions: Drug: Potassium nitrate

INTERVENTIONS:
Drug: Sodium Fluoride — Toothpaste containing 1450 ppm F - EU level as NaF.
  Arms: NaF/KNO3 toothpaste; NaF/KNO3 toothpaste, Low RDA; NaF/KNO3 toothpaste, Medium RDA
Drug: Potassium nitrate — All study treatments contain 5% w/w KNO3.

SUMMARY:
The purpose of this study is to compare and evaluate the ability of two European Union (EU) regulated gel to foam toothpaste formulations versus a non-fluoride toothpaste using a modified in-situ model of dental erosion and remineralization. A positive control i.e fluoride containing toothpaste marketed in EU will also be compared to non-fluoride toothpaste.

DETAILED DESCRIPTION:
The aim of this study is to assess the remineralization effects of two EU gel to foam toothpaste formulations with 1450 parts per million (ppm) of fluoride as sodium fluoride (NaF) and 5% potassium nitrate (KNO3) versus a non-fluoride (0 ppm F)/KNO3 toothpaste as a negative control. The two experimental gel to foam toothpaste formulations differ in their relative dentine abrasivity (RDA) values which is an in-vitro measure of a toothpaste abrasivity to the dentinal tissues. A marketed toothpaste containing NaF and KNO3 will serve as a positive control.

ELIGIBILITY:
Inclusion Criteria:

* General and Oral Health: Good general health with (in the opinion of the investigator) no clinically OST and OHT examinations.
* Oral Requirements:

  * An intact maxillary dental arch suitable for the retention of the palatal appliance and an intact mandibular dental arch. Subjects may have fixed bridges replacing missing teeth.
  * A gum base stimulated whole saliva flow rate ≥ 0.8 g/min and an unstimulated whole saliva flow rate ≥ 0.2 g/min.
* Contraception: Women of childbearing potential who are, in the opinion of the investigator, practicing a reliable method of contraception.

Exclusion Criteria:

* Oral Health:

  * Current active caries or periodontal disease that may compromise the study or the health of the subjects.
  * Lesions of the oral cavity that could interfere with the study evaluations, including severe gingivitis, grossly carious lesions, periodontitis and other severe periodontal disease.
* Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Clinical Study/Experimental Medication:

  * Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit
  * Previous participation in this study
* Substance abuse: Recent history (within the last year) of alcohol or other substance abuse.
* Pregnancy: Women who are pregnant or who are intending to become pregnant over the duration of the study
* Breast-feeding: Women who are breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Groups:
- Overall: This was a 4-way crossover study. Participants brushed with 1.5 g of low relative dentine abrasivity (RDA) gel to foam toothpaste (Toothpaste 1) containing 1450 parts per million (ppm) of fluoride (F) as sodium fluoride (NaF) and 5% weight by weight (w/w) potassium nitrate (KNO3); 1.5 g of medium RDA gel to foam toothpaste (Toothpaste 2) containing 1450 ppm F as NaF and 5% w/w KNO3; 1.5 g of Marketed toothpaste (Toothpaste 3) containing 1450 ppm F as NaF and 5% w/w KNO3; and 1.5 g of placebo toothpaste containing no fluoride but 5% w/w KNO3. There was a washout period of 2 days following each treatment session. In this washout period, participants used a non-fluoridated toothpaste to ensure no carry over effect.
Period: Overall Study
Arm/Group | Overall
Started | 56
Received Placebo (No NaF/KNO3)Toothpaste | 56 (One participant was lost to follow up in study period 1)
Received NaF/KNO3 Toothpaste 1 | 55 (One participant withdrew consent in study period 3)
Received NaF/KNO3 Toothpaste 3 | 54
Received NaF/KNO3 Toothpaste 2 | 55
Completed | 54
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were evaluated for baseline parameters.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.7 (13.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Relative Erosion Resistance (RER) of Enamel Specimens Post 4 Hours of Treatment Exposure
Description: Enamel specimens were exposed to dietary erosive challenge and set of five indentations within each specimen was measured. Decrease in the indentation length compared to the baseline indicates hardening of enamel surface. Enamel specimens were exposed to second erosion challenge to determine RER which compared the indentations values of enamel specimens at baseline (B), first erosive (E1) and second erosive challenge (E2). Percent RER was calculated by formula: [(E1-E2)/ (E1-B)]*100. Smaller the negative RER, better is treatment regimen in imparting resistance to enamel.
Time Frame: Baseline, 4 hours post treatment in each treatment period
Population: Per protocol (PP) population: All randomized subjects who had at least one assessment of efficacy and considered unaffected by major protocol deviations, were included in analysis. Due to drop outs, there was difference in number of participants analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage RER
Groups:
- NaF/KNO3 Toothpaste 1: Participants brushed with 1.5 g of low RDA gel to foam toothpaste containing 1450 ppm F as NaF and 5% w/w KNO3.
- NaF/KNO3 Toothpaste 2: Participants brushed with 1.5 g of medium RDA gel to foam toothpaste containing 1450 ppm F as NaF and 5% w/w KNO3.
- NaF/KNO3 Toothpaste 3: Participants brushed with 1.5 g of NaF/KNO3 toothpaste containing 1450 ppm F as NaF and 5% w/w KNO3.
- No Fluoride/KNO3 Toothpaste: Participants brushed with a fluoride free toothpaste (0 ppmF) containing only 5% w/w KNO3.
Arm/Group | NaF/KNO3 Toothpaste 1 | NaF/KNO3 Toothpaste 2 | NaF/KNO3 Toothpaste 3 | No Fluoride/KNO3 Toothpaste
Number analyzed (Participants) | 55 | 54 | 54 | 56
Percentage RER | -36.66 (2.824) | -36.53 (2.848) | -36.98 (2.847) | -77.82 (2.799)
Statistical Analysis 1: Comparison: NaF/KNO3 Toothpaste 1 vs No Fluoride/KNO3 Toothpaste; Null hypothesis considered population means for the treatments in comparison to be equal with respect to %RER. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 41.15, 95% CI 2-sided [34.42 to 47.89] — Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: NaF/KNO3 Toothpaste 2 vs No Fluoride/KNO3 Toothpaste; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 41.28, 95% CI 2-sided [34.51 to 48.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF/KNO3 Toothpaste 3 vs No Fluoride/KNO3 Toothpaste; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 40.83, 95% CI 2-sided [34.06 to 47.61] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Surface Microhardness (SMH) Recovery of Enamel Specimens Post 4 Hours of Treatment Exposure
Description: SMH test was used to assess mineralization status of enamel specimens using a Wilson 2100 Hardness tester. SMH was determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents rehardening of enamel surface. Percent SMH recovery was calculated from indentation values of enamel specimens at baseline (B), after in-situ hardening (R) and after first erosive challenge (E1) using formula: [(E1- R)/ (E1-B)]*100. A higher percentage values indicate a better outcome.
Time Frame: Baseline, 4 hours post treatment in each treatment period
Population: PP population: All randomized subjects who had at least one assessment of efficacy and considered unaffected by major protocol deviations, were included in analysis. Due to drop outs, there was difference in number of participants analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage SMH
Groups:
- No Fluoride/KNO3 Toothpaste: Participants brushed with a fluoride free toothpaste (0 ppm F) containing only 5% w/w KNO3.
Arm/Group | NaF/KNO3 Toothpaste 1 | NaF/KNO3 Toothpaste 2 | NaF/KNO3 Toothpaste 3 | No Fluoride/KNO3 Toothpaste
Number analyzed (Participants) | 55 | 54 | 54 | 56
Percentage SMH | 32.24 (1.469) | 32.32 (1.480) | 34.53 (1.480) | 22.87 (1.457)
Statistical Analysis 1: Comparison: NaF/KNO3 Toothpaste 1 vs No Fluoride/KNO3 Toothpaste; Null hypothesis considered population means for the treatments in comparison to be equal with respect to %SMH recovery. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 9.36, 95% CI 2-sided [6.01 to 12.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF/KNO3 Toothpaste 2 vs No Fluoride/KNO3 Toothpaste; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 9.45, 95% CI 2-sided [6.07 to 12.82] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF/KNO3 Toothpaste 3 vs No Fluoride/KNO3 Toothpaste; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 11.66, 95% CI 2-sided [8.28 to 15.03] — [estimate comment as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: RER of Enamel Specimens Post 2 Hours of Treatment Exposure
Description: as for outcome 1
Time Frame: Baseline, 2 hours post treatment in each treatment period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: % RER
Arm/Group | NaF/KNO3 Toothpaste 1 | NaF/KNO3 Toothpaste 2 | NaF/KNO3 Toothpaste 3 | No Fluoride/KNO3 Toothpaste
Number analyzed (Participants) | 55 | 54 | 54 | 56
% RER | -43.76 (3.182) | -43.33 (3.211) | -41.88 (3.210) | -85.88 (3.154)

4. Other Pre Specified Outcome: SMH Recovery of Enamel Specimens Post 2 Hours of Treatment Exposure
Description: as for outcome 2
Time Frame: Baseline, 2 hours post treatment in each treatment period
Population: PP population: All randomized subjects who had at least one assessment of efficacy and considered unaffected by major protocol deviations, were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage SMH
Arm/Group | NaF/KNO3 Toothpaste 1 | NaF/KNO3 Toothpaste 2 | NaF/KNO3 Toothpaste 3 | No Fluoride/KNO3 Toothpaste
Number analyzed (Participants) | 55 | 54 | 54 | 56
Percentage SMH | 28.96 (1.600) | 28.92 (1.615) | 28.30 (1.615) | 17.90 (1.585)

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Groups:
- NaF/KNO3 Toothpaste 1: Participants brushed with 1.5 g of low RDA gel to foam toothpaste containing 1450 parts per million of fluoride as NaF and 5% w/w KNO3.
Arm/Group | NaF/KNO3 Toothpaste 1 | NaF/KNO3 Toothpaste 2 | NaF/KNO3 Toothpaste 3 | No Fluoride/KNO3 Toothpaste
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/54 | 0/56
Other Adverse Events (participants affected / at risk) | 2/55 | 0/55 | 1/54 | 2/56
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaF/KNO3 Toothpaste 1 (N=55) | NaF/KNO3 Toothpaste 2 (N=55) | NaF/KNO3 Toothpaste 3 (N=54) | No Fluoride/KNO3 Toothpaste (N=56)
Gingival Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.